CLINICAL TRIAL: NCT01998217
Title: Combination of Remifentanil and Flurbiprofen in Sedation and Analgesia for ESWL of Pancreatic Stone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Jia-feng Wang, M.D., Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rem-ESWL-Pancreas
Record Dates: First submitted 2013-11-19; First posted 2013-11-28 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Pancreatic Stone Disease
Keywords: extracorporeal shock wave lithotripsy; remifentanil; flurbiprofen; pancreatic stone
MeSH Terms: interventions — Remifentanil; Flurbiprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rem group (Active Comparator): Patients in this group receive single infusion of remifentanil with target concentration infusion.
  Interventions: Drug: Remifentanil
- Flur group (Experimental): Patients in this group receive both infusion of flurbiprofen and remifentanil
  Interventions: Drug: Flurbiprofen and remifentanil

INTERVENTIONS:
Drug: Remifentanil — Patients in Rem group receive sedation and analgesia with remifentanil, dose of which will be determined by the up-and-down method.
  Arms: Rem group
Drug: Flurbiprofen and remifentanil — Patients in this group receive sedation and analgesia with flurbiprofen and remifentanil, dose of which was determined by the up-and-down method.
  Arms: Flur group

SUMMARY:
Extracorporeal shock wave lithotripsy (ESWL) of pancreatic stones has been described as an effective approach for stone drainage and pain relief, and general or epidural anesthesia has been reported for such procedure. Single infusion of remifentanil has been described in ESWL of urinary stones, but it has never been described in ESWL of pancreatic stones. Moreover, single infusion of remifentanil might induce several complications, such as postoperative nausea and vomiting. The investigators attended to investigated whether combination of flurbiprofen with remifentanil reduced remifentanil dose and attenuated the complications.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-65 years
* ASA I-II
* ESWL indication was met

Exclusion Criteria:

* patients with hypertension
* patients compromised in cardiopulmonary function
* patients undergoing ESWL for the second or more times

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Visual analogue score of pain | During ESWL procedure

SECONDARY OUTCOMES:
Cardiovascular responses including blood pressure and heart rate | During ESWL procedure

OTHER OUTCOMES:
Side effects | within 24 hours after ESWL procedure
  The side effects including postoperative nausea and vomiting, as well as pruritus.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, Changhai Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Yang YG, Hu LH, Chen H, Li B, Fan XH, Li JB, Wang JF, Deng XM. Target-controlled infusion of remifentanil with or without flurbiprofen axetil in sedation for extracorporeal shock wave lithotripsy of pancreatic stones: a prospective, open-label, randomized controlled trial. BMC Anesthesiol. 2015 Nov 7;15:161. doi: 10.1186/s12871-015-0141-6. PMID 26547293